CLINICAL TRIAL: NCT04270604
Title: Biological Sample Collection for Research and Biobanking
Status: Terminated | Type: Observational
Why Stopped: The study was voluntarily terminated by the PI to focus efforts on an alternative biobanking protocol.
Sponsor: New York Stem Cell Foundation Research Institute (Other)
Responsible Party: Principal Investigator, Laura Andres-Martin, Senior Research Investigator, New York Stem Cell Foundation Research Institute
Other Study IDs: 10-005; 20112091 (Other: WCG IRB)
Record Dates: First submitted 2019-12-20; First posted 2020-02-17 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Parkinson Disease; Diabetes Mellitus, Type 1; Macular Degeneration; ALS; Cancer; Alzheimer Disease; Huntington Disease
Keywords: stem cell; observational; biobank; disease modeling; genetics
MeSH Terms: conditions — Parkinson Disease; Diabetes Mellitus, Type 1; Macular Degeneration; Neoplasms; Alzheimer Disease; Huntington Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Skin biopsy (2-3mm) and/or blood (up to 50 mL); saliva; excess/leftover biospecimens that were (or will be) collected for other purposes (e.g., medical procedure)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Biological sample collection — Biological sample collection for biobanking and research

SUMMARY:
The New York Stem Cell Foundation (NYSCF) Research Institute is performing this research to study different conditions and diseases by using cells from the body (such as skin or blood cells). NYSCF uses these samples to make stem cells and other types of cells, conduct research on the samples, perform genetic testing, and/or store these samples for future use.

Through this research, scientists hope to identify future treatments or even cures.

DETAILED DESCRIPTION:
Researchers at NYSCF study diverse diseases, conditions, and traits by creating "pluripotent" stem cells. These stem cells can become any cell in the human body, including cells that may be difficult, invasive, or even impossible to obtain directly. For example, researchers may create pancreatic insulin-producing cells to learn more about type 1 diabetes, or brain cells to learn more about Parkinson's disease.

Additionally, researchers perform genetic testing to learn more about DNA, a material in most cells that contains instructions for the body's development and functions (such as traits like eye color and risk of certain diseases). A piece of DNA that determines the specific role of a cell is called a "gene." If the instructions in a gene are abnormal, this can lead to disease.

Participation in the study involves: (1) completion of a health questionnaire, (2) providing a skin and/or blood sample from which stem cells may be created, (3) possible collection of a saliva sample for genetic analysis, and (4) possible future follow-up to provide additional information or learn about other research studies.

This study is not a clinical trial.

ELIGIBILITY:
Inclusion Criteria:

Age

* 18 years or older or
* Minor with parent/guardian consent

Biological Sample Collection

* Able and willing to provide:

  * new samples of blood, skin, and/or saliva specifically for use in this study and/or
  * excess/leftover samples, cell lines, and/or derivatives that were (or will be) collected for reasons other than this study

Exclusion Criteria:

* Non-English speaking
* Wards of the state
* For skin samples collected specifically for this study: history of keloid formation, bleeding disorder, allergy to the anesthetic, or anticoagulation use that precludes sample collection.
* For blood samples collected specifically for this study: bleeding disorder, or other medical condition, if the subject's condition increases the risks associated with blood collection.
* For saliva samples: inability to produce sufficient saliva or has a condition that precludes sample collection (such as severe trismus).
* For prospective samples: refuse to adhere to NYSCF's and/or collaborating site's COVID-19 safety protocols during the COVID-19 pandemic.

Ages: 1 Month to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with a diagnosis of one or more of the listed conditions.
  Individuals with a known genetic mutation, with or without a diagnosed condition.
  Individuals without a genetic mutation or condition to serve as healthy controls (a comparison group for those with conditions).
Sampling Method: Non-Probability Sample
Enrollment: 1279 (Actual)
Dates: Start 2012-02-06 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
Establishment of a diverse bank of biological samples, stem cell lines, derivatives, and associated information. | Baseline
  There are no primary endpoints planned for this biobank; endpoints will be specific to research projects that utilize samples/data contained in the biobank. Projects may investigate the biology, etiology, manifestations, progression, risk factors, genetic underpinnings, and treatment of diseases, conditions, and traits.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Andres-Martin, Principal Investigator — New York Stem Cell Foundation Research Institute
Locations (1):
- New York Stem Cell Foundation Research Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: New York Stem Cell Foundation Website — http://nyscf.org